CLINICAL TRIAL: NCT05193201
Title: A Multicenter Phase Ib Clinical Study for Recombinant Human Thrombopoietin Injection in the Treatment of Thrombocytopenia in Patients With Chronic Liver Disease
Brief Title: A Phase Ib Clinical Study for rhTPO in the Treatment of Thrombocytopenia in Patients With Chronic Liver Disease
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenyang Sunshine Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3SBio-TPO-106-Ib-01
Record Dates: First submitted 2021-12-31; First posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Liver Disease Chronic; Thrombocytopenia
Keywords: recombinant human thrombopoietin injection; Thrombocytopenia; Liver Disease Chronic
MeSH Terms: conditions — Thrombocytopenia | interventions — Thrombopoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 : 50*10^9/L ≤ Baseline of PLT < 75*10^9/L (Experimental): The multiple-dose regimen (15000 U subcutaneous injection once a day for 7 days) of recombinant human thrombopoietin (rhTPO) injection for the treatment of thrombocytopenia in patients with chronic liver disease.
  Interventions: Drug: recombinant human thrombopoietin injection
- Cohort 2 : 30*10^9/L ≤ Baseline of PLT < 50*10^9/L. (Experimental): The multiple-dose regimen (15000 U subcutaneous injection once a day for 7 days) of recombinant human thrombopoietin (rhTPO) injection for the treatment of thrombocytopenia in patients with chronic liver disease.
  Interventions: Drug: recombinant human thrombopoietin injection

INTERVENTIONS:
Drug: recombinant human thrombopoietin injection — recombinant human thrombopoietin: 15000 U subcutaneous injection once a day for 7 days
  Other Names: rhTPO

SUMMARY:
The purpose of this study is to explore the multiple-dose regimen of recombinant human thrombopoietin (rhTPO) injection for the treatment of thrombocytopenia in patients with chronic liver disease.

DETAILED DESCRIPTION:
This is a multi-center, open label, phase Ib clinical study. The effectiveness of the multiple-dose regimen of recombinant human thrombopoietin injection in the treatment of thrombocytopenia in patients with chronic liver disease is mainly verified by evaluating the proportion of responders with platelet count in the first 8 days after treatment. Cohort 1 (n=18) : 50*10^9/L ≤ Baseline of PLT < 75*10^9/L. Cohort 2 (n=36) : 30*10^9/L ≤ Baseline of PLT < 50*10^9/L.

ELIGIBILITY:
Inclusion Criteria:

* Gender: There is no limit to men and women.
* 18 years old to 75 years old.
* Liver cirrhosis diagnosed by biopsy/imaging due to chronic liver disease, and Child-Pugh classification is A and B. Patients with liver cirrhosis diagnosed by transient elastography technology can also be included in the group.
* Baseline platelet level: 30×10^9/L≤platelet count<75×10^9/L.
* Liver function ALT and aspartate aminotransferase (AST)≤5×ULN, total bilirubin≤1.5×ULN, blood creatinine≤1.5×ULN.
* Able to understand and be willing to comply with the requirements of the clinical trial protocol, and voluntarily sign a written informed consent form.

Exclusion Criteria:

* Those who are known to be allergic to any component of this product.
* Patients with liver cirrhosis caused by drug-induced liver damage.
* Those with a history of splenectomy or liver transplantation.
* Previously or currently suffering from serious diseases of any organ or system other than the liver, including cardiovascular disease, blood system disease, and nervous system disease patients, as well as any other diseases judged by the investigator to be unsuitable for participating in this trial.
* Currently suffering from malignant tumors, including solid tumors and hematological malignancies.
* Those who are clearly diagnosed as liver failure.
* Liver cirrhosis with serious complications, including: hepatic encephalopathy, refractory ascites, upper gastrointestinal bleeding, etc.;.
* People who have previously or are currently suffering from any disease that may lead to reduced platelet count and/or abnormal platelet function except for chronic liver disease and cirrhosis, including aplastic anemia, myelodysplastic syndrome, myelofibrosis, etc.
* Those who have undergone intrahepatic portosystemic shunt via jugular vein in the past.
* Doppler ultrasound, computerized tomography (CT) or magnetic resonance imaging (MRI) and other imaging examinations that indicate the presence of portal vein thrombosis within 28 days before administration.
* Use heparin, warfarin, non-steroidal anti-inflammatory drugs, aspirin, verapamil, and ticlopidine or glycoprotein IIb/IIIa antagonist (such as tirofiban) within 7 days before administration treat.
* Interferon has been used within 14 days before administration.
* Have received platelet transfusion or used platelet-containing blood products within 14 days before administration, except for transfusion of concentrated red blood cells.
* Those who have received any platelet-increasing therapy within 28 days before administration (the platelet-increasing function of Li Kejun, caffeic acid tablets and/or certain Chinese medicines or Chinese patent medicines that have the function of increasing platelet function can be accepted within 14 days), including but not Limited to rhTPO.
* No more than 28 days after the cessation of other research drug treatments or device research treatments carried out before the administration.
* There are currently patients with WHO ≥ Grade 2 active bleeding, or those with active bleeding in the past 2 weeks.
* Known human immunodeficiency virus positive or Treponema pallidum antibody positive.
* Combined with severe infections that cannot be effectively controlled (except for chronic hepatitis B and chronic hepatitis C).
* The subjects did not agree to take effective contraceptive measures during the trial period. The female subjects had a positive blood pregnancy test during the screening period; women who were pregnant or breastfeeding or had pregnancy plans within 3 months.
* Subjects' understanding, communication and cooperation are not enough to guarantee that the research will be carried out in accordance with the protocol.
* The researcher believes that the subjects are not suitable to participate in this study due to other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-01-16 (Estimated); Primary Completion 2022-10-16 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
the proportion of responders with platelet count | Up to 8 days
  Based on the results of routine blood tests, calculate the proportion of responders with platelet counts in the first 8 days after treatment

SECONDARY OUTCOMES:
the proportion of responders with platelet count | Up to 36 days
  Based on the results of routine blood tests, calculate the proportion of responders with platelet counts during the study
Platelet count | Up to 36 days
  Based on the results of routine blood tests, calculate the change in platelet count from baseline at different visit times after treatment. Calculate the duration of alleviation of thrombocytopenia symptom relief to different levels (≥50×10^9/L; ≥75×10^9/L; ≥100×10^9/L).
Platelet peak | Up to 36 days
  Based on the results of routine blood tests, observe the peak value of platelets and record the peak time after treatment.
AE | Up to 36 days
  All adverse events related to rhTPO observed through various tests (including blood routine, liver function, pregnancy test, electrocardiogram, etc.)
Immunogenicity of rhTPO | At Day 1, Day 14, Day 36
  Detect the presence of anti-rhTPO antibodies through the subject's blood sample
Cmax | Up to 36 days
  Detect the blood concentration of rhTPO by the subject's blood sample
AUC | Up to 36 days
  Detect the blood concentration of rhTPO by the subject's blood sample, then calculate the area under the curve (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Yimin Cui, PhD, Principal Investigator — Peking University First Hospital; Xiaoyuan Lin, Master, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No